CLINICAL TRIAL: NCT03038776
Title: A Randomised, Controlled, Phase 1 Study in Healthy Adults to Evaluate the Immunogenicity and Safety of a Recombinant H7 Hemagglutinin Influenza Vaccine
Brief Title: Recombinant H7 Hemagglutinin Influenza Vaccine Trial
Acronym: FLU007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLU007
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Influenza, Avian
Keywords: vaccine
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Two i.m. administrations 4 weeks apart of recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7 antigen)
  Interventions: Biological: Recombinant influenza hemagglutinin
- 2 (Experimental): Two i.m. administrations 4 weeks apart of recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7 antigen) + Advax-1 adjuvant
  Interventions: Biological: Recombinant influenza hemagglutinin
- 3 (Experimental): Two i.m. administrations 4 weeks apart of recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7 antigen) + Advax-2 adjuvant
  Interventions: Biological: Recombinant influenza hemagglutinin
- 4 (Experimental): Two i.m. administrations 4 weeks apart of T cell epitope modified recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7m antigen) antigen
  Interventions: Biological: Recombinant influenza hemagglutinin
- 5 (Experimental): Two i.m. administrations 4 weeks apart of T cell epitope modified recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7m antigen) + Advax-1 adjuvant
  Interventions: Biological: Recombinant influenza hemagglutinin
- 6 (Experimental): Two i.m. administrations 4 weeks apart of T cell epitope modified recombinant influenza hemagglutinin corresponding to avian H7N9 virus strain (rH7m antigen) + Advax-2 adjuvant
  Interventions: Biological: Recombinant influenza hemagglutinin

INTERVENTIONS:
Biological: Recombinant influenza hemagglutinin — Avian H7N9 influenza vaccine
  Other Names: Panblok-H7

SUMMARY:
Recombinant H7 (rH7) vaccine has been shown to be poorly immunogenic in previous human clinical trials. This study will test approaches to improve the immunogenicity of H7 vaccine, namely use of a three dose regimen, use of a modified H7 HA sequence from which the Tregitope has been removed (rH7m), and inclusion of delta inulin adjuvant adjuvant in the vaccine

DETAILED DESCRIPTION:
Because antibody responses to experimental H7 vaccine have been low even with high antigen doses, there is a need to find ways to enhance the effectiveness of H7 vaccines. Protein Sciences Corporation (PSC) produces an FDA approved seasonal recombinant trivalent influenza vaccine consisting of influenza hemagglutinin proteins (HA) which are full length uncleaved glycoproteins (rHA0) produced using baculovirus expression vectors in cultured insect cells grown in serum-free media (FluBlok®). The mechanism of action of FluBlok is the same as that of traditional inactivated seasonal influenza vaccines.

PanBlok H7 is a pandemic influenza vaccine produced by PSC in the same way as Flublok but it is directed against H7 rather than seasonal influenza virus strains. The vaccine candidate consists of a full-length recombinant monovalent hemagglutinin (rHA) derived from H7N9 virus, in a sterile solution for intramuscular injection. PanBlok H7 rHA is manufactured using the same production process as previously used for Panblok H1/2009pdm ("swine flu") and Panblok H5 pandemic vaccines, both of which vaccines have been previously successfully trialled by us in clinical protocols, FLU005 and FLU003. In both these trials the Panblok antigen was combined with Advax adjuvant formulations. In the FLU005 trial of Panblok H1N1/2009pdm vaccine, the inclusion of Advax adjuvant doubled the seroconversion rate of the vaccine and provided major antigen-sparing effects (Gordon et al, 2012). Whilst the FLU003 trial is ongoing, preliminary data again shows the importance of the Advax adjuvants to vaccine effectiveness. This provides a strong rationale for inclusion of Advax adjuvants in the Panblok H7 vaccine.

It has also been recently recognised that at least one of the reasons for the low immunogenicity of H7 vaccines in human trials to date is that the H7 antigen from this virus contains a T-cell regulatory epitope (Tregitope) in the HA stem region which suppresses the immune response to the vaccine. It was recently demonstrated in humanised animal studies undertaken by collaborators in Japan that removing this Tregitope by modifying 3 amino acids in the H7 stem was able to significantly increase the ability of the H7 vaccine to induce antibody production by human immune cells. This trial will provide the first opportunity to confirm this approach is able to enhance the immunogenicity of H7 in humans, which if confirmed would represent a major breakthough in pandemic influenza vaccine design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years or over
* Able to provide written informed consent
* Willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* History of serious vaccine allergy*
* History of vasculitis, Wegener's granulomatosis, narcolepsy, Guillain Barre, SLE or other systemic autoimmune disease that in the opinion of the investigator would make the vaccine contraindicated
* History of chronic liver disease or liver transaminases elevated more than 3xULN
* Women of childbearing potential, unless using a reliable and appropriate contraceptive method, specifically oral contraceptive pill, IUD or mechanical barrier device.
* Pregnant or lactating women.
* Any serious medical, social or mental condition which, in the opinion of the investigator, would be detrimental to the subjects or the study.
* Receipt of another investigational agent within 28 days preceding initiation of treatment.

  * Individuals who have a past history of potential vaccine reactions will be assessed by the investigator, who will decide whether any past potential vaccine-related side are sufficiently minimal to allow vaccine administration to proceed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Seroconversion | 1 month post immunization
Seroprotection | 1 month post immunization
Fold rise in geometric mean titer | 1 month post immunization

SECONDARY OUTCOMES:
Safety: Frequency and severity of adverse events | 12 months post immunization
  Frequency and severity of adverse events
T cell response | 1 month post-immunization
  Frequency of influenza specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MD, PhD, Principal Investigator — Flinders University/ARASMI
Locations (1):
- Flinders University, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No